CLINICAL TRIAL: NCT02396862
Title: A Prospective, International, Longitudinal, Observational Disease Registry of Patient-reported Outcomes (PROs) and the Association With Hemophilia A and Its Treatment in Patients With Moderate to Severe Hemophilia A
Brief Title: Patient Functioning and Well-being, Economic, and Clinical Impact of Hemophilia A and Its Treatment
Acronym: ECHO
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 17285; KG1301 (Other: Company internal)
Record Dates: First submitted 2015-03-19; First posted 2015-03-24 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; BAY 14-2222

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with moderate to severe Hemophilia A / Cohort 1: Patients aged over 16 years, with documented physician-confirmed diagnosis of moderate or severe Hemophilia A (severity defined as moderate = FVIII activity 1% to 5% and severe = FVIII activity ≤1%)
  Interventions: Drug: Available Recombinant, and Human Factor VIII products incl. Kogenate FS (Recombinant Factor VIII, BAY14-2222)

INTERVENTIONS:
Drug: Available Recombinant, and Human Factor VIII products incl. Kogenate FS (Recombinant Factor VIII, BAY14-2222) — Recombinant and Human Factor VIII / Used on demand or prophylaxis of bleeds

SUMMARY:
The purpose of the study is to improve the understanding of key patient reported outcomes such as quality of life as well as clinical outcomes in hemophilia A, in a global real world setting.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 or over.
* Have documentation of physician-confirmed diagnosis of moderate or severe Hemophilia A (severity defined as moderate = FVIII activity 1% to 5% and severe = FVIII activity ≤1%).
* Signed written informed consent provided by the patient or the patient's parents for patients under the age of 18 (dependent of local regulations).
* Signed written assent is also required for patients under the age 18 years (dependent on local regulations).
* Plan to receive at least half of their Hemophilia care at the registry site.
* Willing and able to enter data as per the data collection schedule.
* Currently receiving prophylactic or on demand treatment (including within last 6months for on demand).
* Expected life expectancy of at least 2 years.

Exclusion Criteria:

* Patients with Hemophilia B
* Patients with von Willebrand disease (vWD)
* Patients with other rare bleeding disorders
* Unable to comply with the study protocol

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged over 16 years, with documented physician-confirmed diagnosis of moderate or severe Hemophilia A (severity defined as moderate = FVIII activity 1% to 5% and severe = FVIII activity ≤1%)
Sampling Method: Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2015-12-09 (Actual); Primary Completion 2018-01-17 (Actual); Study Completion 2018-03-26 (Actual)

PRIMARY OUTCOMES:
Patient Reported Outcome: Change of function as measured by Hemophilia Activities List (HAL), Daily Activities including Work Productivity and Activity Impairment Scale (WPAI). | Baseline and at 12 months
Patient Reported Outcome: Change of function as measured by Hemophilia Activities List (HAL), Daily Activities including Work Productivity and Activity Impairment Scale (WPAI). | Baseline and at 24 months
Patient Reported Outcome: Change of function as measured by Hemophilia Activities List (HAL), Daily Activities including Work Productivity and Activity Impairment Scale (WPAI). | Baseline and at 36 months
Patient Reported Outcome: Change of function as measured by Hemophilia Activities List (HAL), Daily Activities including Work Productivity and Activity Impairment Scale (WPAI). | Baseline and at 48 months
Patient Reported Outcome: Change of function as measured by Hemophilia Activities List (HAL), Daily Activities including Work Productivity and Activity Impairment Scale (WPAI). | Baseline and at 60 months
Patient Reported Outcome: Change of Quality of Life as measured by EuroQol-5 Dimension questionnaire 5 Level (EQ5D), Short Form Health Survey (SF-12), Hemophilia Quality of Life Measure for Adults (HAEMO-QoL-A) | Baseline and at 12 months
Patient Reported Outcome: Change of Quality of Life as measured by EuroQol-5 Dimension questionnaire 5 Level (EQ5D), Short Form Health Survey (SF-12), Hemophilia Quality of Life Measure for Adults (HAEMO-QoL-A) | Baseline and at 24 months
  Resources: Hospital and Healthcare professional visits
Patient Reported Outcome: Change of Quality of Life as measured by EuroQol-5 Dimension questionnaire 5 Level (EQ5D), Short Form Health Survey (SF-12), Hemophilia Quality of Life Measure for Adults (HAEMO-QoL-A) | Baseline and at 36 months
Patient Reported Outcome: Change of Quality of Life as measured by EuroQol-5 Dimension questionnaire 5 Level (EQ5D), Short Form Health Survey (SF-12), Hemophilia Quality of Life Measure for Adults (HAEMO-QoL-A) | Baseline and at 48 months
Patient Reported Outcome: Change of Quality of Life as measured by EuroQol-5 Dimension questionnaire 5 Level (EQ5D), Short Form Health Survey (SF-12), Hemophilia Quality of Life Measure for Adults (HAEMO-QoL-A) | Baseline and at 60 months
Patient Reported Outcome: Change of treatment patterns as measured by Hemophilia Treatment Satisfaction Questionnaire (Hemo-SAT) and Validated Hemophilia Regimen Treatment Adherence Scale (Veritas Pro/PRN) | Baseline and at 12 months
Patient Reported Outcome: Change of treatment patterns as measured by Hemophilia Treatment Satisfaction Questionnaire (Hemo-SAT) and Validated Hemophilia Regimen Treatment Adherence Scale (Veritas Pro/PRN) | Baseline and at 24 months
Patient Reported Outcome: Change of treatment patterns as measured by Hemophilia Treatment Satisfaction Questionnaire (Hemo-SAT) and Validated Hemophilia Regimen Treatment Adherence Scale (Veritas Pro/PRN) | Baseline and at 36 months
Patient Reported Outcome: Change of treatment patterns as measured by Hemophilia Treatment Satisfaction Questionnaire (Hemo-SAT) and Validated Hemophilia Regimen Treatment Adherence Scale (Veritas Pro/PRN) | Baseline and at 48 months
Patient Reported Outcome: Change of treatment patterns as measured by Hemophilia Treatment Satisfaction Questionnaire (Hemo-SAT) and Validated Hemophilia Regimen Treatment Adherence Scale (Veritas Pro/PRN) | Baseline and at 60 months
Patient Reported outcome: Change of adherence as measured by and Validated Hemophilia Regimen Treatment Adherence Scale (Veritas Pro/PRN) | Baseline and at 12 months
Patient Reported outcome: Change of adherence as measured by and Validated Hemophilia Regimen Treatment Adherence Scale (Veritas Pro/PRN) | Baseline and at 24 months
Patient Reported outcome: Change of adherence as measured by and Validated Hemophilia Regimen Treatment Adherence Scale (Veritas Pro/PRN) | Baseline and at 36 months
Patient Reported outcome: Change of adherence as measured by and Validated Hemophilia Regimen Treatment Adherence Scale (Veritas Pro/PRN) | Baseline and at 48 months
Patient Reported outcome: Change of adherence as measured by and Validated Hemophilia Regimen Treatment Adherence Scale (Veritas Pro/PRN) | Baseline and at 60 months
Patient Reported outcome: Change of satisfaction as measured by Hemophilia Treatment Satisfaction Questionnaire (Hemo-SAT) | Baseline and at 12 months
Patient Reported outcome: Change of satisfaction as measured by Hemophilia Treatment Satisfaction Questionnaire (Hemo-SAT) | Baseline and at 24 months
Patient Reported outcome: Change of satisfaction as measured by Hemophilia Treatment Satisfaction Questionnaire (Hemo-SAT) | Baseline and at 36 months
Patient Reported outcome: Change of satisfaction as measured by Hemophilia Treatment Satisfaction Questionnaire (Hemo-SAT) | Baseline and at 48 months
Patient Reported outcome: Change of satisfaction as measured by Hemophilia Treatment Satisfaction Questionnaire (Hemo-SAT) | Baseline and at 60 months
Patient Reported outcome: Change of pain as measured by Brief Pain Inventory (Short Form) (BPI-SF) | Baseline and at 12 months
Patient Reported outcome: Change of pain as measured by Brief Pain Inventory (BPI-SF) | Baseline and at 24 months
Patient Reported outcome: Change of pain as measured by Brief Pain Inventory (BPI-SF) | Baseline and at 36 months
Patient Reported outcome: Change of pain as measured by Brief Pain Inventory (BPI-SF) | Baseline and at 48 months
Patient Reported outcome: Change of pain as measured by Brief Pain Inventory (BPI-SF) | Baseline and at 60 months
Patient Reported outcome: Change of number of resource utilization as evaluated from the patient perspective | Baseline and at 12 months
Patient Reported outcome: Change of number of resource utilization as evaluated from the patient perspective | Baseline and at 24 months
Patient Reported outcome: Change of number of resource utilization as evaluated from the patient perspective | Baseline and at 36 months
Patient Reported outcome: Change of number of resource utilization as evaluated from the patient perspective | Baseline and at 48 months
Patient Reported outcome: Change of number of resource utilization as evaluated from the patient perspective | Baseline and at 60 months
Patient Reported outcome: Change of well-being as measured by Psychological General Well Being Schedule (PGWBI) as well as Smoking and drinking behavior and recreational drug use | Baseline and at 12 months
Patient Reported outcome: Change of well-being as measured by Psychological General Well Being Schedule (PGWBI) as well as Smoking and drinking behavior and recreational drug use | Baseline and at 24 months
Patient Reported outcome: Change of well-being as measured by Psychological General Well Being Schedule (PGWBI) as well as Smoking and drinking behavior and recreational drug use | Baseline and at 36 months
Patient Reported outcome: Change of well-being as measured by Psychological General Well Being Schedule (PGWBI) as well as Smoking and drinking behavior and recreational drug use | Baseline and at 48 months
Patient Reported outcome: Change of well-being as measured by Psychological General Well Being Schedule (PGWBI) as well as Smoking and drinking behavior and recreational drug use | Baseline and at 60 months

SECONDARY OUTCOMES:
Clinical Outcome: Change of Hemophilia A status | Baseline and every 12 months up to 60 months
  Hemophilia A status as defined by: - Last measured FVIII level - History of intracranial hemorrhage and age of occurrence - Number of Bleeding episodes/events in the last year - Location of bleed - Confirmed microbleeds on past imaging - PK assessment (if available): Name of FVIII product for most recent PK evaluation - Dose of Factor VIII product administered for most recent PK evaluation - Measured Factor VIII level - Factor VIII half-life and time point of measurement -- Central Venous Access Device (CVAD) or AV (arterial-venous) fistulae
Clinical Outcome: Change of Joint Status | Baseline and every 12 months up to 60 months
  Joint Status as defined by: - Hemophilia Joint Health Score/ Pettersson Additive Scale - Range of motion - Imaging (where available) - Target joints and past surgical procedures
Clinical Outcome: Baseline disease characteristics | Baseline
  Baseline disease characteristics and disease course as defined by: - Date of diagnosis of Hemophilia A - Age at first treatment with factor replacement therapy (child/adult) - Type of factor VIII gene mutation (if available) - Factor VIII level at initial diagnosis (if available) - History of inhibitor and assay used for detection - Date of determination of peak level of inhibitor
Clinical Outcome: Change of treatment patterns including Hemophilia treatments via patient chart | Baseline and every 12 months up to 60 months
  Treatment patterns as measured by: - Treatment choice and dose (Factor VIII use and type) - Treatment Regimen - Immune tolerance therapy - Products for inhibitors - Blood bank products - Non plasma and topical products

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (10):
- United States (7):
  - Phoenix, Arizona
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - New Orleans, Louisiana
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Columbus, Ohio
- Multiple Locations, Japan
- Multiple Locations, Spain
- Multiple Locations, United Kingdom